CLINICAL TRIAL: NCT03763903
Title: Comparison of 3D Versus 2D Training of Basic Laparoscopic Skills in Terms of Training Effectiveness
Brief Title: Comparison of the Effectiveness of 2D Versus 3D Basic Laparoscopic Skills Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Heinrich Husslein, Assoc.-Prof. Priv.-Doz. Dr., PLL.M., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018_123
Record Dates: First submitted 2018-11-28; First posted 2018-12-04 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Laparoscopy
Keywords: skills training; laparoscopic surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D training (Other): Basic laparoscopic skills (FLS tasks) training using 3D visualization
  Interventions: Other: 3D training
- 2D training (Other): Basic laparoscopic skills (FLS tasks) training using 2D visualization
  Interventions: Other: 2D training

INTERVENTIONS:
Other: 3D training — Skills (FLS tasks) training using 3D visualization
  Arms: 3D training
Other: 2D training — Skills (FLS tasks) training using 2D visualization
  Arms: 2D training

SUMMARY:
The aim of this study is to find out whether basic laparoscopic skills training (FLS tasks) on a standard pelvic trainer using conventional 2D visualization is at least equally effective in terms of skills improvement compared to practicing with 3D visualization. Furthermore, the progress in basic laparoscopic skills improvement for each visualization modality will be analyzed.

DETAILED DESCRIPTION:
An increasing number of operations are done minimal invasively. For example, appendectomy, cholecystectomy, bariatric procedures, colorectal resections as well as hysterectomy and many other gynecologic procedures, are routinely performed laparoscopically.

Laparoscopy requires psychomotor skills that may be difficult to learn and result in prolonged learning curves. In order to become familiar with the 2-dimensional visualization and to learn and improve laparoscopic skills, training is needed. As traditional training in the operating room is expensive and comprises an increased operating risk for the patient, various training alternatives outside the operating room have been developed and shown to be effective in translating the thereby acquired skills to the operating room. Besides training on live animals or cadavers, there are virtual reality simulators, augmented reality simulators and different box trainers. Each of these training devices has specific advantages and limitations. However, some types could be superior to others in terms of training effectiveness. For instance, with implementation of 3D visualization during laparoscopic interventions which facilitates spatial perception, the question arises as to whether training of basic laparoscopic skills using conventional 2D visualization is at least equally effective compared to training with 3D visualization.

The aim of this study is to find out whether basic laparoscopic skills (FLS tasks) training on a standard pelvic trainer using conventional 2D visualization is at least equally effective in terms of skills improvement compared to practicing with 3D visualization. Furthermore, the progress in basic laparoscopic skills improvement for each visualization modality will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* medical students with limited experience in laparoscopic surgery

Exclusion Criteria:

* any laparoscopic operation performed as the primary surgeon
* regular (e.g., once per month) practice on a box trainer for the last 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
Improvement in total Fundamentals of Laparoscopic Surgery (FLS) manual skills scores using 2D versus 3D training of basic laparoscopic skills (using four different FLS tasks) | 5 weeks
  Performance of four different Fundamentals of Laparoscopic Surgery (FLS) tasks will be assessed according to the time needed to complete the task as well as the accuracy of task performance using the FLS scoring system as previously described [Derossis AM, Fried GM, Abrahamowicz M, et al. Development of a model for training and evaluation of laparoscopic skills. Am J Surg 1998;175:482-7.]. The improvement of performance for the total score as well as for each FLS task will be calculated by subtracting the baseline test scores from the posttraining test scores. The primary outcome measure will be the improvement in total test scores.

SECONDARY OUTCOMES:
Progress in basic laparoscopic skills improvement according to the time required for completion of the different FLS tasks during the training period in the 3D and the 2D visualization group | 5 weeks
  Analysis of the progress in basic laparoscopic skills improvement according to the time required for FLS task completion during the training period for each of the two visualization modalities

CONTACTS AND LOCATIONS:
Overall Officials: Heinrich Husslein, MD, PLL.M., Principal Investigator — Department of Obstetrics and Gynecology, Medical University of Vienna
Locations (1):
- Medical University Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No